CLINICAL TRIAL: NCT05398744
Title: MIGHTEE: Motivational Interviewing and Group Heart Transplant Exercise and Education: A Pilot Study
Brief Title: Motivational Interviewing and Group Heart Transplant Exercise and Education: A Pilot Study
Acronym: MIGHTEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-018888
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Orthotopic Heart Transplant
Keywords: OHT; Aerobic Exercise; Motivational interviewing; Group Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual group aerobic training program (Experimental): 16-week, virtual group aerobic training program led by exercise physiologist. Duration: 24 weeks. Four weeks recording of baseline activity through activity monitor; 16-week virtual group aerobic training program, 3 times per week for 30 minutes; and four weeks of follow-up.
  Interventions: Other: Group Exercise Program

INTERVENTIONS:
Other: Group Exercise Program — At-home, aerobic group exercise program facilitated by exercise physiologist via video format, 3 times a week for 16 weeks.

SUMMARY:
The aim of this 16-week group aerobic training program, delivered remotely via video-conferencing, is to assess program feasibility, and determine if program increases physical activity in adolescents after heart transplant.

DETAILED DESCRIPTION:
Orthotopic heart transplant (OHT) is the definitive therapy for children with cardiac disease, however, survival after transplant is limited, and quality of life after transplant is less than healthy peers'. The transplanted heart usually works well, pumping blood as well as most healthy hearts. As such, the American Heart Association recommends no specific exercise related restrictions for heart transplant recipients. Although most children have normal cardiac function after OHT, children with transplanted hearts have impaired exercise performance, and do not exercise as much as their peers. This finding is concerning, as impaired exercise tolerance is associated with reduced survival, diminished health related quality of life, and depression and anxiety. These factors negatively impact adherence, and further limit graft survival. Thus, identifying interventions that positively impact physical activity and promote graft longevity, like individualized exercise programs, should be a priority for post-transplant care.

Investigators propose that increasing physical activity in children and adolescents after OHT may be a critical modifiable method for increasing graft longevity and improving quality of life. Investigators will explore this through a pilot program. Participants will wear an activity monitor to record physical activity, parents/caregivers and participants will complete surveys, and participants will engage with psychologists and exercise physiologists.

ELIGIBILITY:
Inclusion Criteria for Patients

* Age 12-18 years old
* More than 12 months removed from their initial heart transplant
* Agreement to participate in study protocol and willing/able to return for follow-up.
* Access to computer and/or internet for uploading health data from wearable electronic activity monitor.
* Access to an electronic device (phone, tablet, or computer) with a camera feature, microphone, and the capacity to use Zoom, the virtual platform which will stream the group exercise session.
* Clinical EKG with normal sinus rhythm
* English language proficiency

Exclusion Criteria for Patients

* Patients who are restricted from exercise
* Patients who are pregnant
* History of pharmaceutically treated rejection within the prior 6 months
* Physical or behavioral conditions that would prevent them from participating in aerobic exercise (i.e., significant motor disability, illness precluding participation in the exercise regimen as described).
* Inability to complete a standard maximal exercise stress test (as defined by those who did not achieve an respiratory exchange ratio (RER)>1.1 and who gave submaximal effort according to exercise physiologist performing EST)
* EKG or ambulatory rhythm monitor performed within the last 12 months which shows 2nd or 3rd degree atrioventricular (AV) block
* Patients with a medication change after their baseline EST expected to affect their heart rate response to exercise (i.e. initiation/discontinuation of a beta-blocker, beta-agonist during exercise, or ivabradine)
* Pacemaker

Inclusion Criteria for Parents

* Parent of a patient that fits all inclusionary/exclusionary eligibility criteria
* English language proficiency at least at a 5th grade level or for limited English proficient (LEP) parents, preferred language proficiency of at least a 5th grade level

Exclusion Criteria for Parents

- Unwilling to complete questionnaires

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Study feasibility assessed by participation in training sessions | 16 weeks
  Attendance at assigned training sessions
Study feasibility evaluated by participants' engagement on the activity monitor application | 24 weeks
  Days of logged activity on the MyHeart application
Study feasibility assessed by participants' engagement with exercise physiologist | 24 weeks
  Participants' attendance at biweekly meetings with exercise physiologist

SECONDARY OUTCOMES:
Physical activity of participants | 24 weeks
  Time spent at target heart rate
Health Related Quality of life | 24 weeks
  Health related quality of life (HRQL) will be measured by participants' responses to Pediatric Quality of Life (PEDSQL) questionnaire, generating scores from 0-100 with a higher score indicating better quality of life.
Psychological well-being | 24 weeks
  Psychological well-being will be evaluated by participants' responses on questionnaires using Patient Reported Outcome Measurement Information System (PROMIS). PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population (usually U.S. general population) with a higher score indicating more of the psychological concept being measured.
Perceived exercise barriers or exercise barriers | 24 weeks
  Exercise barriers will be measured by analysis of survey responses related to physical activity practices
Participants' overall program satisfaction | 24 weeks
  Participants' overall program satisfaction will be analyzed by review of completed post-intervention questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Edelson, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No